CLINICAL TRIAL: NCT00082277
Title: A Multicentre Phase III/IV Study, of the Effects of Risedronate Sodium (ACTONEL™, 35mg/Week, Oral) on Bone, in Postmenopausal Women, With Hormone-receptor-positive Early Breast Cancer, Treated With Anastrozole (ARIMIDEX™, 1mg/Day Oral) With Risk of Fragility Fracture (High-risk Fragility Fracture-open-label, Non-comparative Stratum; Moderate-risk of Fragility Fracture-randomised, Double-blind Stratum; Low-risk of Fragility Fracture - Open-label, Non-comparative Stratum)Abbreviated
Brief Title: Anastrozole Biphosphonate Study in Postmenopausal Women With Hormone-Receptor-Positive Early Breast Cancer
Acronym: SABRE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Francisco Sapunar, MD - Arimidex Medical Science Director, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D5392C00050; SABRE
Record Dates: First submitted 2004-05-05; First posted 2004-05-06 (Estimated); Last update posted 2011-01-26 (Estimated); Status verified 2011-01

CONDITIONS: Breast Cancer
Keywords: hormone-receptor positive, breast cancer; Osteopenia; Osteoporosis; risk of fracture; bone loss
MeSH Terms: conditions — Breast Neoplasms; Bone Diseases, Metabolic; Osteoporosis | interventions — Anastrozole; Risedronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- 1 (Experimental): High-Risk Fragility Fracture-Open-Label, Non-Comparative Stratum
  Interventions: Drug: Anastrozole; Drug: Risedronate Sodium
- 2 (Experimental): Moderate-Risk of Fragility Fracture-Randomised, Double-Blind Stratum
  Interventions: Drug: Anastrozole; Drug: Risedronate Sodium
- 3 (Experimental): Low-Risk of Fragility Fracture - Open-Label, Non-Comparative Stratum
  Interventions: Drug: Anastrozole; Drug: Risedronate Sodium

INTERVENTIONS:
Drug: Anastrozole — 1mg/Day Oral
  Other Names: ARIMIDEX™; ZD1033
Drug: Risedronate Sodium — 35mg/week, oral
  Other Names: ACTONEL™

SUMMARY:
The purpose of this study is to evaluate safety parameters of anastrozole with regard to its potential effects on postmenopausal bone loss and on lipid profiles. This trial is conducted to investigate the effects of risedronate on BMD and on bone metabolism in postmenopausal women using anastrozole as adjuvant therapy for hormone-receptor-positive early breast cancer and who are high or moderate risk of fragility fracture. It is also conducted to determine the effects of anastrozole on bone mineral density (BMD) and on bone metabolism in women at low risk of fragility fracture.

ELIGIBILITY:
Inclusion Criteria:

* Women defined as Postmenopausal
* Histologically proven operable invasive breast cancer
* Hormone-receptor-positive breast cancer

Exclusion Criteria:

* Clinical evidence of metastatic disease
* Bilateral hip fractures or bilateral hip prosthesis
* Receiving or received in last 12 months hormonal therapy for breast cancer, bisphosphonate therapy, oestrogens
* Malabsorption syndrome

Min Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2004-04; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
The change from baseline in lumbar spine (L1-L4) bone mineral density (BMD) | Assessed at 12 months

SECONDARY OUTCOMES:
Change from baseline in total hip BMD | Assessed at 12 and 24 months
Change from baseline in lumbar spine (L1-L4) BMD | Assessed at 24 months
Change from baseline in bone formation markers | Assessed at 6 and12 months
Change from baseline in bone resorption and formation markers | Assessed at 6 and 12 months
Change from baseline in LDL-cholesterol | Assessed at 12 months
Change from baseline in LDL-cholesterol, HDL-cholesterol, total cholesterol, and serum triglycerides | Assessed at 3, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Arimidex Medical Science Director, MD, Study Director — AstraZeneca
Locations (35):
- United States (8):
  - Research Site, Palm Springs, California
  - Research Site, Jacksonville, Florida
  - Research Site, New Orleans, Louisiana
  - Research Site, New York, New York
  - Research Site, Raleigh, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Houston, Texas
- Canada (5):
  - Research Site, Burnaby
  - Research Site, Edmonton
  - Research Site, Montreal
  - Research Site, Québec
  - Research Site, Vancouver
- France (5):
  - Research Site, Bordeaux
  - Research Site, Caen
  - Research Site, Lyon
  - Research Site, Saint-Cloud
  - Research Site, Saint-Herblain
- Greece (2):
  - Research Site, Athens
  - Research Site, Irakleio
- Netherlands (4):
  - Research Site, Goes
  - Research Site, Ijssel
  - Research Site, Nijmegen
  - Research Site, The Hague
- South Africa (3):
  - Research Site, Bloemfontain
  - Research Site, Cape Town
  - Research Site, Tygerberg
- Spain (4):
  - Research Site, Pamplona
  - Research Site, Pontevedra
  - Research Site, Seville
  - Research Site, Valencia
- United Kingdom (4):
  - Research Site, Belfast
  - Research Site, Bolton
  - Research Site, Dundee
  - Research Site, Luton

REFERENCES:
- [Derived] Adams A, Jakob T, Huth A, Monsef I, Ernst M, Kopp M, Caro-Valenzuela J, Wockel A, Skoetz N. Bone-modifying agents for reducing bone loss in women with early and locally advanced breast cancer: a network meta-analysis. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD013451. doi: 10.1002/14651858.CD013451.pub2. PMID 38979716